CLINICAL TRIAL: NCT06503965
Title: Design and Rationale of the National Multicenter Tunisian Registry of Trans Catheter Aortic Valve Implantation Registry
Brief Title: Tunisian Registry of Trans Catheter Aortic Valve Implantation
Acronym: TAVI-TN
Status: Recruiting | Type: Observational
Sponsor: Les Laboratoires des Médicaments Stériles (Industry)
Collaborators: Tunisian Society of Cardiology and Cardiovascular Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: TAVI-TN
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-07

CONDITIONS: Tunisian Patients Already Implanted With a TAVI
Keywords: TAVI; Death; Vascular complications; Pacemaker implantation; Echocardiography
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Transcatheter aortic valve implantation (TAVI) has emerged as a transformative therapy for patients with severe aortic stenosis, particularly those designated high-risk or inoperable for traditional surgical valve replacement. Despite its increasing adoption worldwide, there re-mains a paucity of data regarding TAVI outcomes in Tunisian patients. In response to this gap in knowledge, the investigators propose the establishment of the Tunisian TAVI Registry, a multicenter initiative aimed at comprehensively documenting the clinical characteristics, procedural de-tails, and short- and long-term outcomes of TAVI procedures across Tunisia. The TAVI.TN registry will enroll consecutive patients undergoing TAVI procedures at participating centers across Tunisia, between 2013 and 2024 with a retrospective arm and a prospective arm. The TAVI-TN Registry represents a significant step towards enhancing our understanding of TAVI outcomes in the Tunisian population. By systematically capturing real-world data, this initiative aims to inform clinical decision-making, improve patient care, and contribute to the advancement of TAVI practices in Tunisia and beyond.

ELIGIBILITY:
Inclusion Criteria:

- Any Tunisian patient who was treated with TAVI implantation in Tunisia

Exclusion Criteria:

* Patients who are not Tunisians
* Patients not agreeing to sign consent, witnesses not agreeing to sign consent (family member)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * All Tunisian patients already implanted with a TAVI
  * Patients implanted during the period of one year starting from D1 of the registry's launch i.e. 23/09/2023.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-09-23 (Actual); Primary Completion 2025-06-23 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
VARC (Valve Academic Research Consortium-2) defined "Clinical Efficacy" composite endpoint | From 30 days post procedure to completion of at least 2 years of follow up
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Requiring hospitalizations for valve-related symptoms or worsening congestive heart failure
  * NYHA (New York Heart Association) class III or IV functional classification of heart failure
  * Valve-related dysfunction (mean aortic valve gradient ≥20 mmHg, Effective Orifice Area (EOA) ≤0.9-1.1 cm2(c) and/or Doppler Velocity Integral (DVI) <0. 35 m/s, AND/OR moderate or severe prosthetic valve regurgitation

SECONDARY OUTCOMES:
VARC defined 'Device success' composite endpoint | 30 days
  * Absence of procedural mortality
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location
  * Intended performance of the prosthetic heart valve (no prosthesis - patient mismatch and mean aortic valve gradient ,20 mmHg or peak velocity ,3 m/s, no moderate or severe prosthetic valve regurgitation)

CONTACTS AND LOCATIONS:
Overall Officials: Nadhem HAJLAOUI, PI, Principal Investigator — Hôpital militaire principal d'instruction de Tunis
Locations (1):
- Hôpital militaire principal d'instruction de Tunis, Tunis, Tunisia

REFERENCES:
- [Background] Carroll JD, Mack MJ, Vemulapalli S, Herrmann HC, Gleason TG, Hanzel G, Deeb GM, Thourani VH, Cohen DJ, Desai N, Kirtane AJ, Fitzgerald S, Michaels J, Krohn C, Masoudi FA, Brindis RG, Bavaria JE. STS-ACC TVT Registry of Transcatheter Aortic Valve Replacement. Ann Thorac Surg. 2021 Feb;111(2):701-722. doi: 10.1016/j.athoracsur.2020.09.002. Epub 2020 Nov 16. PMID 33213826
- [Background] Alasnag M, AlMerri K, Almoghairi A, Alenezi A, Bardooli F, Al-Sheikh S, Alanazi N, AlHarbi W, Al Lawati H, Al Faraidy K, AlShehri M, Thabane M, Thabane L, Al-Shaibi K. One-Year Outcomes for Patients Undergoing Transcatheter Aortic Valve Replacement: The Gulf TAVR Registry. Cardiovasc Revasc Med. 2022 Aug;41:19-26. doi: 10.1016/j.carrev.2021.12.024. Epub 2021 Dec 31. PMID 35033460
- [Background] Didier R, Le Breton H, Eltchaninoff H, Cayla G, Commeau P, Collet JP, Cuisset T, Dumonteil N, Verhoye JP, Beurtheret S, Lefevre T, Iung B, Gilard M; STOP-AS, France-TAVI investigators. Evolution of TAVI patients and techniques over the past decade: The French TAVI registries. Arch Cardiovasc Dis. 2022 Apr;115(4):206-213. doi: 10.1016/j.acvd.2022.04.004. Epub 2022 Apr 27. PMID 35527212
- [Background] Tezuka T, Higuchi R, Hagiya K, Saji M, Takamisawa I, Nanasato M, Iguchi N, Shimizu A, Shimizu J, Doi S, Okazaki S, Sato K, Tamura H, Yokoyama H, Onishi T, Tobaru T, Takanashi S, Takayama M. Midterm Outcomes of Underweight Patients Undergoing Transcatheter Aortic Valve Implantation: Insight From the LAPLACE-TAVR Registry. JACC Asia. 2022 Dec 13;3(1):78-89. doi: 10.1016/j.jacasi.2022.08.014. eCollection 2023 Feb. PMID 36873767
- [Background] Ciardetti N, Ciatti F, Nardi G, Di Muro FM, Demola P, Sottili E, Stolcova M, Ristalli F, Mattesini A, Meucci F, Di Mario C. Advancements in Transcatheter Aortic Valve Implantation: A Focused Update. Medicina (Kaunas). 2021 Jul 14;57(7):711. doi: 10.3390/medicina57070711. PMID 34356992